CLINICAL TRIAL: NCT01568931
Title: Local Delivery of thrombolytIcs Before Thrombectomy in patientS With ST-elevatiOn myocardiaL Infarction Undergoing Primary percuTaneous Coronary interventION - The DISSOLUTION Randomized Trial
Brief Title: Local Thrombolytics Before Thrombectomy in STEMI
Acronym: DISSOLUTION
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Pelliccia, Assistant Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 197/2012/D
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Coronary Artery Disease
Keywords: thrombectomy
MeSH Terms: conditions — Coronary Artery Disease | interventions — Urokinase-Type Plasminogen Activator; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Urokinase (Active Comparator): Patients will be randomized to to receive local bolus of 200,000 units urokinase
  Interventions: Drug: Urokinase
- Saline (Active Comparator): Patients will be randomized to to receive local bolus of intracoronary saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Urokinase — intracoronary, urokinase, 200,000 Units, bolus
  Other Names: UROKINASE-R, IMARX THERAPEUTICS INC., Tucson, AZ
  Arms: Urokinase
Drug: Saline — intracoronary, saline, bolus 1 cc
  Other Names: Saline infusion
  Arms: Saline

SUMMARY:
Background Prompt reperfusion with percutaneous coronary intervention (PCI) in the setting of ST-elevation myocardial infarction (STEMI) improves clinical outcomes through salvage of myocardial tissue.

Although the use of thrombus aspiration with PCI can result in improved rates of normal epicardial flow and myocardial perfusion, several unmet needs remain.

Purpose The purpose of this trial will be to evaluate the hypothesis that local delivery of thrombolytics vs. saline infusion prior to thrombus aspiration and PCI is safe and effective in patients with STEMI.

DETAILED DESCRIPTION:
The study will select patients with ST-elevation myocardial infarction (STEMI) with angiographic evidence of massive thrombosis in the culprit artery undergoing manual thrombectomy followed by primary percutaneous coronary intervention (PCI).

Patients will be randomized to receive local bolus of 200,000 units urokinase or saline solution

ELIGIBILITY:
Inclusion Criteria:

* ST-elevation myocardial infarction
* angiographic evidence of massive thrombosis in the culprit artery
* Indication to manual thrombectomy followed by primary percutaneous coronary intervention (PCI)
* Able to understand and willing to sign the informed CF

Exclusion Criteria:

* Women of child bearing potential patients must demonstrate a negative pregnancy test performed within 24 hours before CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2020-03 (Actual); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Outcomes at 30 days | Up to 30 days
  30-day occurrence of death, new Q-wave myocardial infarction, coronary artery bypass grafting, target lesion revascularization, stroke, or stent thrombosis

SECONDARY OUTCOMES:
Myocardial reperfusion after Primary CI | Up to 90 minutes after Primary PCI
  ST-segment resolution (STR)>70% as assessed 90 minutes after Primary PCI
Left ventricular remodeling | Up to 1 year after Primary PCI
  A change in left ventricular end-diastolic volume>20% (compared with baseline values) as assessed at 1-year echocardiography
5-year MACE | Up to 5 years after Primary PCI
  Death, reinfarction, new-onset severe heart failure, and rehospitalization for heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Cesare Greco, MD, Study Director — University Sapienza